CLINICAL TRIAL: NCT03418168
Title: An Open-label, Multicenter Study to Investigate the Efficacy and Safety of Oral Molidustat in Peritoneal Dialysis Subjects With Renal Anemia
Brief Title: A Study of Molidustat for Treatment of Renal Anemia in Peritoneal Dialysis Subjects
Acronym: MIYABI PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19353
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anemia; Renal Insufficiency, Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molidustat (BAY85-3934) (Experimental): Molidustat group
  Interventions: Drug: Molidustat (BAY85-3934)

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — Starting dose of molidustat once daily (OD) will be titrated based on the subject's Hb (Hemoglobin) response

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of molidustat in peritoneal dialysis subjects with renal anemia

ELIGIBILITY:
Inclusion Criteria:

* Subject with end-stage kidney disease (ESKD) on peritoneal dialysis prior to assignment and not expected to start maintenance dialysis (e.g., hemodialysis, hemodiafiltration) other than peritoneal dialysis during the study period
* Body weight > 40 and ≤ 160 kg at screening
* Male or female subject ≥ 20 years of age at screening
* At least one kidney
* Subjects who meet one of the 1 or 2 following criteria

  * Subjects untreated with ESA at assignment: Mean of the last 2 Hb level (central laboratory measurement) during the screening period must be ≥ 8.0 and < 11.0 g/dL (2 measurements must be taken ≥ 2 days apart and the difference between the 2 measurements must be < 1.2 g/dL) with the last screening Hb measurement within 14 days prior to study drug assignment
  * Subjects pre treated with ESA at assignment: Mean of the last 2 Hb level (central laboratory measurement) during the screening period must be ≥ 10.0 and < 13.0 g/dL (2 measurements must be taken ≥ 2 days apart and the difference between the 2 measurements must be < 1.2 g/dL) with the last screening Hb measurement within 14 days prior to study drug assignment
* Subjects who meet one of the 1 or 2 following criteria

  * Subjects untreated with ESA at assignment: Subject with ESKD on peritoneal dialysis for at least 2 weeks prior to assignment. AND. Subject not received ESA for 8 weeks prior to assignment. OR. In case of the patient washed out from ESAs, when mean of the last 2 Hb level (at least 2 central laboratory measurements must be taken ≥ 2 days apart) has decrease to ≥ 0.5g/dL from the Hb level (central laboratory measurement) after the last ESA administration, AND the interval from the last ESA administration to the study drug assignment should be over 2 week for epoetin-alpha/beta, 4 weeks for darbepoetin alpha or epoetin beta pegol
  * Subjects pre treated with ESA at assignment:

    * Subject with ESKD on peritoneal dialysis for at least 12 weeks prior to assignment
    * Subject treated with ESA by IV or SC within 8 weeks prior to assignment
    * Treated with 2 or 4 weekly dose of darbepoetin alfa, 4 weekly dose of epoetin beta pegol, OR 3 times per week, twice per week, weekly or bi-weekly dose of epoetin alfa/beta, and having had no more than one dose change within 8 weeks prior to assignment

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, pulmonary thromboembolism, and acute limb ischemia) within 6 months prior to randomization
* Sustained and poorly controlled arterial hypertension (defined as systolic BP≥ 180mmHg or diastolic BP ≥ 110mmHg) or hypotension (defined as systolic BP < 90mmHg) at randomization
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy requiring invasive treatment (e.g., intraocular injections or laser photocoagulation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Responder rate: proportion of responders among the subjects | Week 30 to 36
  Responder is defined as meeting all of the following criteria:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment

SECONDARY OUTCOMES:
Mean Hb (Hemoglobin) level | Week 30 to 36
Change in mean Hb level | Baseline and Week 30 to 36
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 8 weeks
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 4 weeks
Proportion of subjects who meet each component of the response | Week 30 to 36
  Response:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Hb level | Baseline and Up to Week 36
Change in Hb level | Baseline and Up to Week 36
Proportion of subjects with mean hemoglobin levels are in the target range | Week 30 to 36
Proportion of subjects with mean hemoglobin levels are above the target range | Week 30 to 36
Proportion of subjects with mean hemoglobin levels are below the target range | Week 30 to 36
Proportion of subjects with hemoglobin levels in the target range | Up to 36 weeks
Proportion of subjects with hemoglobin levels above the target range | Up to 36 weeks
Proportion of subjects with hemoglobin levels below the target range | Up to 36 weeks
Proportion of subjects whose maximum rise in Hb between each consecutive visits is above 0.5 g/dL/week | Up to 36 weeks
  Defined as change in Hb level / duration between two visits (weeks)
Percentage of days in the target Hb range during the evaluation period | Week 30 to 36
Percentage of days in the target Hb range during the treatment period | Up to 36 weeks
Rate of rise in Hb level (g/dL/week) between each consecutive visits | Up to 36 weeks
Percentage of Hb levels in target range during the evaluation period | Week 30 to 36
  Defined as the number of measurements in the target range / number of measurements x 100 [%])
Percentage of Hb levels in target range during the treatment period | Up to 36 weeks
  Defined as the number of measurements in the target range / number of measurements x 100 [%])
Proportion of subjects who received at least one rescue treatment | Up to 36 weeks
Proportion of subjects whose Hb level was ≥ 13.0 g/dL or < 8.0 g/dL | Up to 36 weeks
Number of participants with serious adverse events | Up to 36 weeks
Maximum concentration (Cmax) of Molidustat | Baseline, Week 8, Wee16 and Week 36
Area under the concentration-time curve (AUC) of Molidustat | Baseline, Week 8, Wee16 and Week 36
EPO (Erythropoietin) serum concentration of Molidustat | Baseline, Week 8, Wee16 and Week 36

CONTACTS AND LOCATIONS:
Locations (27):
- Japan (27):
  - Kainan Hospital, Yatomi, Aichi-ken
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - JCHO Kyushu Hospital, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Elm Grove Clinic, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Toranomon Hospital Kajigaya, Kawasaki, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Niigata Prefectural Shibata Hospital, Shibata, Niigata
  - National Hospital Organization Beppu Medical Center, Beppu, Oita Prefecture
  - Okinawa prefectural Chubu Hospital, Uruma, Okinawa
  - Fuchu Hospital, Izumi, Osaka
  - Fukui-ken Saiseikai Hospital, Fukui
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Asahi University Hospital, Gifu
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Nara Prefecture General Medical Center, Nara
  - Niigata City General Hospital, Niigata
  - Osaka General Medical Center, Osaka
  - Japanese Red Cross Oita Hospital, Ōita

REFERENCES:
- [Derived] Akizawa T, Taguchi M, Matsuda Y, Iekushi K, Yamada T, Yamamoto H. Molidustat for the treatment of renal anaemia in patients with dialysis-dependent chronic kidney disease: design and rationale of three phase III studies. BMJ Open. 2019 Jun 14;9(6):e026602. doi: 10.1136/bmjopen-2018-026602. PMID 31203241
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/